CLINICAL TRIAL: NCT05778513
Title: Evaluation of Endothelial and Vascular Functions in Obese Patients: Analysis of the Blood Flow in the Femoral Artery During Passive Movements of the Limbs
Brief Title: Evaluation of Endothelial and Vascular Functions in Obese Patients (FUENVASOB)
Acronym: FUENVASOB
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C122
Record Dates: First submitted 2023-02-27; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Obesity
Keywords: Obesity; Endothelial function; Vascular function; Passive leg movements
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples

GROUPS / COHORTS (2):
- Cases: Male subjects with obesity
  Interventions: Other: Passive knee flexion-extension + Cycle ergometer exercise + 3-week body weight reduction program
- Controls: Male subjects without obesity
  Interventions: Other: Passive knee flexion-extension + Cycle ergometer exercise

INTERVENTIONS:
Other: Passive knee flexion-extension + Cycle ergometer exercise + 3-week body weight reduction program — Passive knee flexion-extension movements + Incremental cycle ergometer exercise + Multidisciplinary body weight reduction program with a duration of 3 weeks
  Groups: Cases
Other: Passive knee flexion-extension + Cycle ergometer exercise — Passive knee flexion-extension movements + Incremental cycle ergometer exercise
  Groups: Controls

SUMMARY:
The primary objective of the present study will be to evaluate, in obese patients, the blood flow response in the femoral artery in response to passive limb movements, taken as a biomarker of a possible limitation of the peripheral vascular-endothelial-microvascular function. The values will be compared with those obtained in normal subjects, in patients with cardiovascular (Gilford & Richardson 2017) or respiratory diseases (Ives et al. 2020), and in healthy subjects subjected to bed rest (Zuccarelli et al. 2020).

The data of the recruited obese patients will be obtained at the beginning and the end of the standard rehabilitation period (including calorie reduction interventions, physical exercise, and psychological counseling) conducted over 3 weeks at the Division of Auxology, Istituto Auxologico Italiano, Piancavallo, Italy. A secondary objective will be to evaluate any changes following the rehabilitation program on the patients' endothelial-peripheral-vascular-microvascular function. The data obtained will also be evaluated in comparison with hematochemical and molecular indices for evaluating the endothelial function, as well as with standard parameters for the overall functional evaluation of the oxidative function and the ability to sustain exercise ("peak" O2 consumption during exercise, thresholds anaerobic diseases.

DETAILED DESCRIPTION:
Materials and methods:

The study will be attended by 15 young obese males aged between 15 and 40 years recruited at the Division of Auxology (minors) and the Division of Metabolic Diseases (adults), Istituto Auxologico Italiano, IRCCS, Piancavallo, Italy.

The inclusion criteria for the study group will be:

1. BMI > 97th percentile for age and gender (minors) and >35 (adults).
2. not having done structured physical activity programs (regular activity for more than 120 min/week) during the 6 months preceding the study.
3. absence of pathologies such as diabetes or insulin resistance.
4. absence of signs/symptoms referable to cardiovascular, respiratory, gastrointestinal or musculoskeletal pathologies contraindicated for carrying out the tests.

Furthermore, 15 male control subjects of similar age, with normal BMI, will be recruited among friends and colleagues from the Department of Medical Area, University of Udine, who will have to satisfy the inclusion criteria 2-4 mentioned above.

The anthropometric characteristics and body composition of the patients will be determined by tetrapolar impedance analysis (Human-IM Scan, DS-Medigroup, Milan, Italy).

Experimental protocols The tests will be conducted under strict medical supervision, following standard safety protocols. The proposed measures are non-invasive, with the exception of venous blood sampling.

At the beginning and at the end of the standard period of stay of the patient at the Hospital (hospitalization/rehabilitation period lasting 3 weeks, including a combined intervention of aerobic physical activity, caloric restriction and psychological counseling), each subject will undergo, on two different days, to the following protocols:

1. On the first day, the blood flow in the common femoral artery will be determined continuously, by Echo-Doppler method (duplex mode) during passive knee flexion-extension movements (passive leg movement, PLM). To perform this measurement, the subject will assume a sitting position on a special seat. After adequate familiarization, the subject will perform two repetitions, lasting about one minute each, separated by a few minutes of intervals, of a series of passive movements (limb guided by an operator) of flexion and extension of a lower limb (width of movement 90°; knee angle 180°-90°-180°), with a frequency of 1 Hz. During passive movements, the blood flow in the common femoral artery will be determined by Echo-Doppler (duplex mode). The blood flow will be calculated, according to standardized procedures and with the synchronization with the ECG tracing, based on the measured values of femoral artery diameter (B-mode) and blood flow velocity (pulse-vawe mode). The data obtained during the two repetitions of the experiment will be superimposed on each other for analysis. From the tracing of the blood flow as a function of time, the following evaluation parameters of the peripheral vascular-microvascular function will be calculated: blood flow peak; difference between peak flow and resting flow; area under the blood flow versus time curve.
2. On the second day, the patient will perform incremental cycle ergometer exercise (3 minutes rest, 20 watts for 2 minutes and then 20 watt/min increments) conducted until voluntary exhaustion, for determination of "peak" O2 consumption (V̇O2 peak) and of the "ventilatory thresholds".

   Lung ventilation, V̇O2 and carbon dioxide emission (V̇CO2) will be determined breath-by-breath by CPX express metabolizer (Medical Graphics Corporation, St Paul, MN, USA). Arterial oxygen saturation (SaO2) will be determined by earlobe pulse oximetry. The heart rate (heart rate [HR]) will be determined on the basis of the electrocardiographic (ECG) signal, while the arterial pressure will be determined by a sphygmomanometer. The perception of fatigue will be determined using a Borg 6-20 scale.
3. Venous blood samples will be collected from the antecubital vein of the arm, before the protocol described in point 1) and immediately after the incremental exercise described in point 2). On the blood samples, evaluation variables of endothelial function and inflammation markers will be determined.

A portion of the sample will be delivered, following specific protocols, to the Analysis Laboratory of the Piancavallo Hospital, where the following variables will be determined:

Total and HDL cholesterol, HOMA-IR (insulinemia, blood glucose), alpha-1 glycoprotein, CRP, IL-6, TNF-alpha, ICAM-1, VCAM-1, testosterone, cortisol, insulin, irisin, pancreatic peptide, GH, plasma lactate; nitrites, nitrates, prostacyclin (6-keto), von Willebrand factor, endothelin, hyaluronic acid, syndecan, heparan sulfate; Plasma and serum BDNF, plasma TrkB receptor; BCAA (leucine, isoleucine, valine) and BCAA (3 hydroxy-isobutyrate) metabolites (valine intermediate).

ELIGIBILITY:
Inclusion Criteria:

* BMI > 97th percentile for age and gender (minors) and >35 (adults).
* not having done structured physical activity programs (regular activity for more than 120 min/week) during the 6 months preceding the study.
* absence of pathologies such as diabetes or insulin resistance.
* absence of signs/symptoms referable to cardiovascular, respiratory, gastrointestinal or musculoskeletal pathologies contraindicated for carrying out the tests.

Exclusion Criteria:

* having done structured physical activity programs (regular activity for more than 120 min/week) during the 6 months preceding the study
* presence of diabetes or insulin resistance
* presence of signs/symptoms referable to cardiovascular, respiratory, gastrointestinal or musculoskeletal pathologies contraindicated for carrying out the tests.

Ages: 15 Years to 40 Years | Sex: Male
Age Groups: Child, Adult
Study Population: Male obese subjects (BMI > 97th percentile for age and gender (minors) and >35 (adults), hospitalized for a multisciplinary integrated 3 week body weight reduction program
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood flow in the femoral artery in Cases | At baseline and at end of test, before and after 3 weeks of body weight reduction program
  Change from baseline in blood flow in the femoral artery to Passive knee flexion-extension + Cycle ergometer exercise
Change from baseline in blood flow in the femoral artery in Controls | At baseline and at end of test
  Change from baseline in blood flow in the femoral artery to Passive knee flexion-extension + Cycle ergometer exercise

SECONDARY OUTCOMES:
Evaluation of variables of endothelial function and inflammation markers - CRP | Baseline and after 3 weeks
  Change in C-reactive Protein concentration
Evaluation of variables of endothelial function and inflammation markers - IL-6 | Baseline and after 3 weeks
  Change in Interleukin-6 concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Site Piancavallo, Oggebbio, Verbania, Italy